CLINICAL TRIAL: NCT02728830
Title: A Pilot Study Investigating the Effect of Pembrolizumab on the Tumoral Immunoprofile of Gynecologic Cancers of Mullerian Origin
Brief Title: A Study of Pembrolizumab on the Tumoral Immunoprofile of Gynecologic Cancers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AA Secord (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, AA Secord, Professor of Obstetrics & Gynecology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00068544
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Gynecologic Neoplasms; Epithelial Ovarian Cancer; Uterine Endometrial Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: gynecologic cancers; mullerian cancers; tumoral immunoprofile
MeSH Terms: conditions — Genital Neoplasms, Female; Carcinoma, Ovarian Epithelial; Endometrial Neoplasms; Fallopian Tube Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab (Experimental): Subjects will receive one dose of 200mg pembrolizumab by IV 14-21 days prior to surgery. Subjects will undergo standard surgical cytoreductive surgery as deemed appropriate by their gynecologic oncologist, followed by standard adjuvant chemotherapy for their cancer as deemed appropriate by their treating physician.
  If subject's disease does not get worse following standard of care chemotherapy, they will receive pembrolizumab in the maintenance setting every three weeks for up to a year.
  If subject's disease returns after completing a year of pembrolizumab and they have not had adverse reactions to pembrolizumab they may be eligible to continue receiving pembrolizumab for an additional year in the second course phase.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg IV
  Other Names: Keytruda

SUMMARY:
The ultimate goal of the study is to identify potential biomarkers, immune gene expression signatures, and co-stimulatory pathways that may be used to understand the effect of immune checkpoint inhibitors on gynecologic cancers.

DETAILED DESCRIPTION:
Epithelial gynecologic malignancies are tumors of müllerian origin, which include ovarian, endometrial, fallopian tube, and primary peritoneal cancers, and account for >70,000 new diagnoses and >22,000 deaths per year in the United States alone. Treatment typically consists of a thorough cytoreductive and staging surgery in combination with platinum/taxane chemotherapy. Newer approaches adding anti-angiogenic therapies to chemotherapy have resulted in moderate improvements in recurrence free survival. However, despite these aggressive treatments, the majority of women with advanced stage at diagnosis will experience relapse. Unfortunately, relapsed disease is incurable and women ultimately die of their disease despite maximal efforts at cancer control using subsequent chemotherapy or targeted agents. There has been significant interest in incorporating immune checkpoint therapies in the treatment of gynecologic malignancies, especially given the durable remissions associated with these therapies in the treatment of melanoma and early indications of durable responses in recurrent ovarian cancer. At this time, little is known about whether or how to combine chemotherapy, anti-angiogenic therapies, and immunologic therapies for maximal benefit. Understanding the tumor microenvironment, particularly immune and angiogenic factors that contribute to tumor survival, as well as the changes that occur in response to immunotherapy is critical to identify favorable biomarker profiles which could lead to improved prognostic outcomes and inform the development and sequencing of therapies to maximize benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed gynecologic tumor of müllerian origin, specifically epithelial ovarian, fallopian tube, primary peritoneal, or uterine endometrial cancer.
2. Have disease amenable to surgical resection.
3. Be willing and able to provide written informed consent for the trial.
4. Be at least 18 years of age on day of signing informed consent.
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement of the investigator.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined below. All screening labs should be performed within 10 days of study drug administration:

7a. ANC ≥ 1,500/mcL

7b. Platelets ≥ 100,000/mcL

7c. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)

7d. Serum creatinine ≤ 1.5 times the upper limit of normal or calculated creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 times institutional upper limit of normal

7e. Serum total bilirubin ≤ 1.5 times the upper limit of normal or direct bilirubin ≤ the upper limit of normal with total bilirubin levels > 1.5 times upper limit of normal

7f. AST and ALT ≤ 2.5 times the upper limit of normal or ≤ 5 times the upper limit of normal for subjects with liver metastases

7g. Albumin > 2.5 mg/dL

7h. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

7i. Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

8. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity until planned hysterectomy/oophorectomy. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria:

1. Is currently participating and receiving a study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the study drug administration.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study drug administration.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has received prior chemotherapy, targeted small molecule therapy, or radiation therapy for the current gynecologic malignancy.

   NOTE: Subjects who have received treatment for a prior unrelated malignancy must have recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   NOTE: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to study drug administration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study drug administration. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 39 subjects that were consented, 24 were screen failures. Nine were screen failures because exclusionary surgery, 6 because of exclusionary pathology, 3 because physician decision, 2 because of participant withdrawals, 1 was lost to follow up, 1 had exclusionary lab values, 1 had a contraindicated illness, and 1 had a language barrier.
Groups:
- Pembrolizumab: Subjects will receive one dose of 200mg pembrolizumab by IV 14-21 days prior to surgery. Subjects will undergo standard surgical cytoreductive surgery as deemed appropriate by their gynecologic oncologist, followed by standard adjuvant chemotherapy for their cancer as deemed appropriate by their treating physician.
  If subject's disease does not get worse following standard of care chemotherapy, they will receive pembrolizumab in the maintenance setting every three weeks for up to a year.
  If subject's disease returns after completing a year of pembrolizumab and they have not had adverse reactions to pembrolizumab they may be eligible to continue receiving pembrolizumab for an additional year in the second course phase.
  Pembrolizumab: Pembrolizumab 200mg IV
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 39
Completed | 15
Not Completed | 24
Not completed — Exclusionary Surgery | 9
Not completed — Exclusionary Pathology | 6
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Exclusionary Lab Values | 1
Not completed — Contraindicated Illness | 1
Not completed — Language Barrier | 1

BASELINE CHARACTERISTICS:
Population: Analysis was conducted only on subjects who completed the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 63.7 [43 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Primary Tumor Site [Count of Participants; unit: Participants]
  Ovary | 9
  Fallopian Tube | 3
  Uterus | 2
  Other | 1
Histologic Subtype [Count of Participants; unit: Participants]
  Adenocarcinoma; serous | 12
  Adenocarcinoma; clear cell | 3
Tumor Grade at Diagnosis [Count of Participants; unit: Participants]
  High Grade | 10
  Low Grade | 2
  Grade Cannot be Assessed | 3
FIGO Stage of Cancer at Diagnosis [Count of Participants; unit: Participants] — This measure is the stage of the cancer as determined by the FIGO (International Federation of Gynecology and Obstetrics) system.
  Stage I is the least severe, where the tumor is restricted to the organ of origin.
  Stage II involves invasion of surrounding organs or tissue. Stage III involves spread to the distant lymph nodes or tissue within the pelvis.
  Stage IV involves distant metastasis beyond the peritoneal cavity.
  Participants
    I | 1
    II | 0
    III | 9
    IV | 1
    Unstaged | 4
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance Status (ECOG) is a way for physicians to track changes in a subject's level of functioning on a 5 point scale. An ECOG score of 0 is a subject who is fully active and able to carry on all pre-disease performance without restriction. An ECOG score of 1 is restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature (e.g. light house work). The higher the score, the more restricted in level of function and capability of self-care
  Participants
    0 | 5
    1 | 10
Debulking Surgery [Count of Participants; unit: Participants] — This measure depicts that amount of residual disease that was left at the time of surgery completion. Optimal R0 notes that no residual disease was left after surgery. Optimal R1 notes that less than 1cm of residual disease remained. Suboptimal debulking notes that macroscopic residual disease was left at the end of surgery.
  Participants
    Optimal R0 | 7
    Optimal R1 | 5
    Suboptimal | 2
    Not Applicable | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Immune Infiltrates as Measured by PD-L1 Modified H-Score
Description: This outcome measures the change in tumor immune infiltrates post-pembrolizumab versus pre-pembrolizumab as measured by the PD-L1 Modified H-score.
  Histological score (H-score) is a score that is comprised of intensity and percentage of staining and is used for assessing amount of protein (in this case PD-L1) present in a tissue sample. H-score is determined by adding of the percentages of cell staining at each intensity level multiplied by the membrane intensity of staining (0 (no staining), 1+ (weak staining), 2+ (medium staining), 3+(strong staining)).
  The H-score has a range of 0 to 300. Lower H-scores represent lower expression of PD-L1 in the tumor sample, while higher scores represent stronger expression of PD-L1 in the tumor samples.
Time Frame: Baseline and 14-21 Days
Population: Eleven subjects had adequate matched pre- and post- treatment tissue samples for analysis for tumor immune infiltrates.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 11
score on a scale | 13.2 (23.2)

2. Secondary Outcome: Toxicity Profile: Frequency and Severity of Adverse Events as Assessed by CTCAE
Description: Frequency and severity of adverse events associated with pembrolizumab when given to patients with newly diagnosed gynecologic cancers of müllerian origin prior to standard surgical therapy and as maintenance therapy after completion of chemotherapy. All events experienced within the AE reporting time frame deemed probably, possibly, or definitely related to study drug above the reporting threshold of 4%. Categorized by grade and frequency, defined using CTCAE 4.0 event name and grading.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 15
Participants
  Anemia, Grade 1 | 2
  Neutropenia, Grade 2 | 1
  Thrombocytopenia, Grade 1 | 2
  Abdominal pain, Grade 1 | 5
  Abdominal pain, Grade 2 | 2
  ALT elevation, Grade 1 | 8
  ALT elevation, Grade 2 | 1
  ALT elevation, Grade 3 | 1
  AST elevation, Grade 1 | 7
  AST elevation, Grade 2 | 1
  AST elevation, Grade 3 | 3
  ALK phosphatase elevation, Grade 1 | 7
  ALK phosphatase elevation, Grade 2 | 1
  Arthralgia, Grade 1 | 3
  Anorexia, Grade 1 | 2
  Anorexia, Grade 2 | 2
  Back pain, Grade 1 | 2
  Bloating, Grade 1 | 1
  Bloating, Grade 2 | 2
  Constipation, Grade 1 | 2
  Constipation, Grade 2 | 2
  Diarrhea, Grade 1 | 6
  Diarrhea, Grade 2 | 9
  Diarrhea, Grade 3 | 2
  Dyspnea, Grade 2 | 2
  Edema, Grade 1 | 3
  Fatigue, Grade 1 | 12
  Fatigue, Grade 2 | 2
  Headache, Grade 1 | 8
  Hypertension, Grade 1 | 1
  Hypertension, Grade 2 | 2
  Hypertension, Grade 3 | 1
  Hypoalbuminemia, Grade 1 | 2
  Hypomagnesemia, Grade 1 | 3
  Hypomagnesemia, Grade 2 | 1
  Hyponatremia, Grade 1 | 3
  Hyponatremia, Grade 3 | 1
  Nausea, Grade 1 | 13
  Nausea, Grade 2 | 4
  Proteinuria, Grade 1 | 1
  Proteinuria, Grade 2 | 2
  Proteinuria, Grade 3 | 1
  Vomiting, Grade 1 | 13
  Weight loss, Grade 1 | 3

3. Other Pre Specified Outcome: Exploratory: Changes in Tumoral and Circulating Blood Immunoprofile
Description: To characterize changes in the tumoral and circulating blood immunoprofile after administration of pembrolizumab. Levels of immune and inflammatory mediators, profile of tumor immune infiltrates, and the expression of PD-L1 in pre-administration samples will be compared to post-administration surgical resection (including ascites) samples.
Time Frame: Baseline and 14-21 Days
Population: Thirteen participants had pre and post samples available for analysis
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 13
fold change
  CXCL10 Fold Change, Pre to Post Pembro | 1.5 [1.4 to 2.0]
  IFN-Gamma Fold Change, Pre to Post Pembro | 1.6 [1.0 to 1.8]
  IL12p70 Fold Change, Pre to Post Pembro: number analyzed (Participants) | 12
  IL12p70 Fold Change, Pre to Post Pembro | 1.1 [0.7 to 1.7]
  IL1b Fold Change, Pre to Post Pembro: number analyzed (Participants) | 11
  IL1b Fold Change, Pre to Post Pembro | 1.9 [0.7 to 3.6]
  IL2ra Fold Change, Pre to Post Pembro | 1.2 [1.0 to 1.4]
  IL6 Fold Change, Pre to Post Pembro | 1.1 [0.9 to 1.3]
  TNF-Alpha Fold Change, Pre to Post Pembro | 1.1 [1.0 to 1.2]

4. Other Pre Specified Outcome: Exploratory: Changes in Tumoral and Circulating Blood Immunoprofile for Those Who Enroll in Second Course Phase at Time of Recurrence
Description: To evaluate changes in the tumoral and circulating blood immunoprofile at time of recurrence. Levels of immune and inflammatory mediators, profile of tumor immune infiltrates, and the expression of PD-L1 in samples at time of recurrence will be compared to pre-administration and surgical samples.
Time Frame: 18 months
Population: No enrolled subjects qualified for the second course phase
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study collected AEs and SAEs from the time of informed consent to 30 days after the first Pembrolizumab infusion, an average of 1 month. AEs and SAEs were also collected during the Pembrolizumab maintenance phase. They were not collected while subjects were receiving standard of care chemotherapy.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=15)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=15)
Anemia (Blood and lymphatic system disorders) | 7
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 5
INR increased (Investigations) | 1
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 5
Fever (General disorders) | 3
General disorders and administration site conditions- Other, specify (General disorders) | 4 — One event: Large ventral hernia One event: Dysuria One event: Right foot drop One event: Swelling abdominal
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Papulopustular rash (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Reproductive system and breast disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders- other, specify (Respiratory, thoracic and mediastinal disorders) | 2 — One event: Bronchitis One event: Shortness of breath
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders- other, specify (Skin and subcutaneous tissue disorders) | 1 — One event: Dry lips
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02728830/Prot_SAP_000.pdf